CLINICAL TRIAL: NCT04067115
Title: SARC037: A Phase I/II Study to Evaluate the Safety of Trabectedin Administered as a 1-Hour Infusion in Ewing Sarcoma Patients in Combination With Low Dose Irinotecan and 3'-Deoxy-3'-18F Fluorothymidine (18F-FLT) Imaging
Brief Title: SARC037: A Phase I/II Study to Evaluate the Safety of Trabectedin in Combination With Irinotecan in Ewing Sarcoma Patients
Acronym: U01CA236220
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SARC037; U01CA236220 (NIH)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Trabectedin; Irinotecan; alovudine; X-Rays

STUDY DESIGN:
Intervention Model Description: This phase I study will follow a standard 3+3 design and the Phase II study will be a single-arm, mini-max Simon two-stage design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trabectedin and Irinotecan (Experimental): Trabectedin will be delivered by infusion on day 1 followed by 2 doses on irinotecan delivered by infusion for one hour on day 2 and day 4 of 21 day cycles. Some patients will receive an 18F-FLT Imaging scan prior to the first administration of trabectedin and once after administration of trabectedin.
  Interventions: Drug: Trabectedin 1 MG [Yondelis]; Drug: Irinotecan; Diagnostic Test: tumor biopsy; Other: 3'-Deoxy-3'-18F Fluorothymidine (18F-FLT) Imaging

INTERVENTIONS:
Drug: Trabectedin 1 MG [Yondelis] — Patients with Ewing sarcoma will be administered trabectedin intravenously. Cycles are 21 days.
Drug: Irinotecan — Patients with Ewing sarcoma will be administered inirotecan intravenously. Cycles are 21 days.
Diagnostic Test: tumor biopsy — Tumor tissue samples will be collected collected at two timepoints. The first biopsy will be prior to treatment. If a biopsy is not possible archival tissue may be submitted. A second tumor biopsy will be taken fro consenting patients when possible after the first administration of Trabectedin to evaluate the effect on the tumor cells.
Other: 3'-Deoxy-3'-18F Fluorothymidine (18F-FLT) Imaging — Some patients will receive PET scans with the use of 18F-FLT, a radioactive tracer, performed at the National Institute of Health.
  Other Names: 18F-FLT Imaging

SUMMARY:
This study evaluates the trabectedin and irinotecan in the treatment of Ewings sarcoma, with a EWS-FLI1 mutation. Patients will also receive an infusion of 18F-FLT in combination with a Positron Emission Tomography (PET) scan to help evaluate the effect of treatment.

DETAILED DESCRIPTION:
Trabectedin and Irinotecan may inhibit the activity of this Ewing sarcoma mutation. Trabectedin may suppress the proliferation of the gene involved in DNA damage response. It blocks EWS-FLI1 by inactivating the fusion protein and silences the target genes.

Irinotecan also suppresses the genes regulating the tumor cells, generating DNA damage. Together, these drugs work in combination to suppress the gene regulating the tumor cells. This combination may suppress the activity of the tumor regulating genes, disrupting the activity of the genes. The infusion of 18F-FLT in combination with a Positron Emission Tomography (PET) scan will demonstrate whether the target cells have been suppressed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsed and refractory Ewing sarcoma with EWS-FLI1 fusion type for which there is no known therapy proving to prolong survival
* measurable disease
* ECOG Performance Status of 0-2 or Lansky of 50
* adequate organ function
* written, voluntary consent
* willing to undergo tumor biopsy
* negative hepatitis infection

Exclusion Criteria:

* prior therapy with trabectedin or lurbinectedin
* known history of hypersensitivity to irinotecan or topotecan or their excipients.
* known brain metastases
* known bleeding diathesis
* pregnant or breastfeeding
* currently receiving other investigational drugs or anticancer agents
* clinically significant unrelated illness or uncontrolled infection
* unable to comply with the safety monitoring requirements

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Phase I The recommended dose (RD) of trabectedin administered in combination with low dose irinotecan | up to 36 months
  The recommended dose will be established by enrolling patients at the lowest dose and observing them for dose limiting toxicity. Dose limiting toxicity describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. The maximum tolerated dose is the highest dose of a drug or treatment that does not cause unacceptable side effects. If 0 of the first 3 subjects experience DLT, the study will proceed to the next dose level. If 1 subject experiences a DLT, that dose level cohort will be expanded to 6 total subjects. If no additional subjects experience DLTs at that dose level cohort, the study will proceed to enroll the next dose level cohort.
  If ≥ 2 of 6 subjects experience DLT, then that dose level is the recommended dose of trabectedin (RD). The study will proceed to the same process for the irinotecan escalation.
  If 2 or all 3 subjects experience DLT, that dose level is the recommended dose of trabectedin (RD).
Phase I Tumor response rate | up to 36 months
  The anti-tumor activity of the combination of trabectedin and low-dose irinotecan as measured by the tumor objective response rate (ORR) assessed by RECIST v1.1
Phase 2 To determine anti-tumor activity of the combination trabectedin and low-dose irinotecan | up to 36 months
  Tumor objective response rate (ORR) assessed by RECIST v1.1.

SECONDARY OUTCOMES:
Phase I/Phase 2 Tumor response rate, progression-free survival (PFS), duration of response, and 6-month PFS rate of patients with ES treated with trabectedin and irinotecan. | up to 36 months
  The percentage of patients whose tumor shrinks or disappears after treatment (per RECIST 1.1), progression-free survival (PFS) of patients with ES treated with trabectedin and irinotecan.
Phase I monitor the avidity of Ewing sarcoma tumors of EWS-FLI1 12-24 hours after trabectedin administration and before irinotecan is administered and before 18F-FLT PET scans | up to 36 months
  18F-FLT PET avidity of Ewing sarcoma tumors.
Phase 2 To determine anti-tumor activity of the combination trabectedin and low-dose irinotecan | up to 36 months
  The anti-tumor activity of the combination of trabectedin and low-dose irinotecan as measured by the tumor objective response rate (ORR) assessed by RECIST v1.1
Phase I/Phase 2 Tumor response rate, progression-free survival (PFS), duration of response, and 6-month PFS rate of patients with ES treated with trabectedin and irinotecan. | up to 36 months
  The percentage of patients whose tumor shrinks or disappears after treatment (per RECIST 1.1) duration of response of patients with ES treated with trabectedin and irinotecan.
Phase I/Phase 2 Tumor response rate, progression-free survival (PFS), duration of response, and 6-month PFS rate of patients with ES treated with trabectedin and irinotecan. | up to 36 months
  The percentage of patients whose tumor shrinks or disappears after treatment (per RECIST 1.1) duration of 6-month PFS rate ES treated with trabectedin and irinotecan.

OTHER OUTCOMES:
Progression free survival | up to 5 years
  The time from starting treatment until disease progression
6- month Progression free survival | up to 36 months
  To determine the rate of disease progression at 6 months after starting treatment
Duration of Response | up to 5 years
  The time from tumor response to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Grohar, MD/PhD, Principal Investigator — Children's Hospital of Philadelphia; John Glod, MD/PhD, Study Director — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - National Cancer Institute, Bethesda, Maryland
  - Boston Children's Hospital / Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania